CLINICAL TRIAL: NCT03914586
Title: The OXIRIS Filter in Septic Shock : the Adsorption of Endotoxin and Cytokines Improves the Haemodynamic , the Renal Function , and the Metabolic Response
Brief Title: The Membrane Adsorbing OXiris Filter in Septic Patients With AKI
Acronym: MOSAKI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: FRANCO TURANI (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor-Investigator, FRANCO TURANI, Adjunt Professor of Anesthesia and Intensive Care, University of Rome Tor Vergata
Organization: University of Rome Tor Vergata (Other)
Other Study IDs: 418/CE Lazio 1
Record Dates: First submitted 2019-04-11; First posted 2019-04-16 (Actual); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Sepsis; Acute Renal Failure
Keywords: Sepsis; Acute Renal Failure; Extra Corporeal Therapy
MeSH Terms: conditions — Sepsis; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Septic patients with AKI: Patients with sepsis /septic shock ( Sepsis III ) and AKI submitted to Continuous Renal Replacement Therapy with the adsorbing membrane oXiris.
  Interventions: Device: oXiris filter

INTERVENTIONS:
Device: oXiris filter — Continuous Renal Replacement Therapy with oXiris filter

SUMMARY:
Patients with Sepsis / Septic Shock and AKI are submitted to Continuous Renal Replacement Therapy with the oXiris filter . The pro- inflammatory mediators , the endotoxin , interleukin 10 , the main cardiorespiratory indices and renal parameters are evaluated at the entry of the study and at the end of the treatment.

DETAILED DESCRIPTION:
Patients with a diagnosis of sepsis or septic shock Gram + , Gram - and acute renal failure All patients are submitted to Continuous Renal Replacement Therapy with the treated heparin-coated membrane (oXiris;Baxter );

* Citrate Anticoagulation or Heparin with thromboelasthograpy monitoring .
* Hemodynamic monitoring with dynamic parameters ( Cardiac Index ,Stroke Volume Variation , Pulse Pressure Variation ) and Echocardiography
* Indirect Calorimetry ( before Continuous Renal Replacement Therapy and after 1 hour stopping Continuous Renal Replacement Therapy )
* Laboratory: white blood cell, creatinine, procalcitonin, Interleukin -6, Interleukin -10, Endotoxin , Lactate, diuresis, tromboelastography (post filter and arterial sample ) and dosage of Plasminogen Activator Inhibitor -1 at the same sites.

ELIGIBILITY:
Inclusion Criteria:- Age <18 years 75 years >

* Diagnosis of sepsis or septic shock (Sepsis III)
* Mechanical Ventilation or non Invasive ventilation with PaO2 /FIO2 < 200.
* Renal failure ( AKI ≥ 1)
* Endotoxin ( EAA ) : EAA ≥ 0.6 -0.9 > or IL6 > 150 pg/mL

Exclusion Criteria:

* Pregnancy;
* Age < 18 years 75>
* Chronic Renal failure or previous CRRT
* Immunological disease or immunosuppressive drugs or EAA < 0.6 with IL 6 in the normal range.
* CGS < 8 due to hemorrhagic or ischemic event.
* ECMO v-v or a-v or ECCO2 removal.
* No resolution of the surgical source of infection
* Terminal condition
* Any contraindication to heparin and other anticoagulant.
* Other pathological conditions in which the oXiris filter is not indicated and other therapeutic options are required. (eg . Hepatic failure , Cardiac failure )

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with sepsis /septic shock and AKI
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-01-10 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
Hemodynamic Data | At the 24 - 48 hours after starting of the treatment
  Changes of vasoactive drugs concentration (micr/Kg/min)
Renal Data | At the 24 - 48 hours after starting of the treatment
  Changes of Urinary Out Put ( mL/ 24 hours)
Respiratory Data | At the 24 - 48 hours after starting of the treatment
  Changes of P/F ratio
Calorimetric data | At the 24 - 48 hours after starting of the treatment
  Changes of VO2 (mL / min)

SECONDARY OUTCOMES:
Inflammatory data | At the 24 - 48 hours after starting of the treatment
  Changes of Endotoxin ( EAA measurement )
Coagulation data | At the 24 - 48 hours after starting of the treatment
  Changes of the PAI-1 ( ng /mL)
Cytokines Data | At the 24 - 48 hours after starting of the treatment
  IL 6 (pg/mL)
Cytokines data | At the 24 - 48 hours after starting of the treatment
  IL 10 (pg/mL)

CONTACTS AND LOCATIONS:
Locations (1):
- Franco Turani, Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Malard B, Lambert C, Kellum JA. In vitro comparison of the adsorption of inflammatory mediators by blood purification devices. Intensive Care Med Exp. 2018 May 4;6(1):12. doi: 10.1186/s40635-018-0177-2. PMID 29728790
- [Background] Turani F, Barchetta R, Falco M, Busatti S, Weltert L. Continuous Renal Replacement Therapy with the Adsorbing Filter oXiris in Septic Patients: A Case Series. Blood Purif. 2019;47 Suppl 3:1-5. doi: 10.1159/000499589. Epub 2019 Apr 12. PMID 30982024